CLINICAL TRIAL: NCT05874557
Title: Effects of Compound Amino Acid Capsule on Nutrition, Calcium and Phosphorus Metabolism in Maintenance Hemodialysis Patients
Brief Title: A Study of Compound Amino Acid Capsule on Maintenance Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2023-0042
Record Dates: First submitted 2023-04-14; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- treatment group: MHD patients who took compound amino acid capsules regularly(2# tid po) for 9 months
- control group: MHD patients in the control group are selected by PSM with age, sex, dialysis month, baseline BMI, baseline Kt/V and baseline ultrafiltration volume. And they did not take compound amino acid capsules or similar amino acid nutritional supplement for the same 9 months.

SUMMARY:
The goal of this retrospective cohort study is to investigate the effects of compound amino acid capsule on nutrition, calcium and phosphorus metabolism in maintenance hemodialysis(MHD) patients. The main questions it aims to answer are:

1. Can compound amino acid capsule improve the nutritional status of MHD patients?
2. Can compound amino acid capsule help to correct the calcium and phosphorus metabolism imbalance of MHD patients?
3. Is compound amino acid capsule safe for MHD patients? We will collect the medical history and laboratory data of MHD patients who regularly took compound amino acid capsule for 9 months or did not use the same preparation in previous medical experience. We focus on the difference of serum albumin level between the treatment group and the control group within 9 months, as well as prealbumin, hemoglobin, ferritin, calcium, phosphorus, 1,25-OH 2-D3 and intact parathyroid hormone (iPTH).

ELIGIBILITY:
Inclusion Criteria:

* Patients who received maintenance hemodialysis (≥ 3 months) in Renji Hospital;
* Regularly participate in the routine laboratory examination of the hemodialysis center every 3 months;
* Inclusion criteria of the treatment group: regular treatment with compound amino acid capsule for 9 months (2 tablets, 3 times a day, orally);
* Inclusion criteria of the control group: no compound amino acid capsules or similar nutritional supplement were taken.

Exclusion Criteria:

* Severe heart failure (NYHA III/IV);
* Human immunodeficiency virus positive or is suffering from other serious infectious diseases;
* Have a history of malignant tumor;
* Women during pregnancy or lactation;
* Exclusion criteria for treatment group: previous use of amino acids or compound ketoacid supplement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: maintenance hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Serum Albumin at 3 months | Data of both groups at baseline and 3 months are collected and analyzed.
  Change from baseline serum albumin at 3 months of the treatment group and control group are compared.
Change from Baseline Serum Albumin at 6 months | Data of both groups at baseline and 6 months are collected and analyzed.
  Change from baseline serum albumin at 6 months of the treatment group and control group are compared.
Change from Baseline Serum Albumin at 9 months | Data of both groups at baseline and 9 months are collected and analyzed.
  Change from baseline serum albumin at 9 months of the treatment group and control group are compared.

SECONDARY OUTCOMES:
Change from Baseline Prealbumin at 3 months of the treatment group | Data of the treatment group at baseline and 3 months are collected and analyzed.
  Within the treatment group, prealbumin at 3 months is compared to baseline. In other words, change from baseline prealbumin at 3 months is compared to 0.
Change from Baseline Prealbumin at 3 months of the control group | Data of the control group at baseline and 3 months are collected and analyzed.
  Within the control group, prealbumin at 3 months is compared to baseline. In other words, change from baseline prealbumin at 3 months is compared to 0.
Change from Baseline Prealbumin at 6 months of the treatment group | Data of the treatment group at baseline and 6 months are collected and analyzed.
  Within the treatment group, prealbumin at 6 months is compared to baseline. In other words, change from baseline prealbumin at 6 months is compared to 0.
Change from Baseline Prealbumin at 6 months of the control group | Data of the control group at baseline and 6 months are collected and analyzed.
  Within the control group, prealbumin at 6 months is compared to baseline. In other words, change from baseline prealbumin at 6 months is compared to 0.
Change from Baseline Prealbumin at 9 months of the treatment group | Data of the treatment group at baseline and 9 months are collected and analyzed.
  Within the treatment group, prealbumin at 9 months is compared to baseline. In other words, change from baseline prealbumin at 9 months is compared to 0.
Change from Baseline Prealbumin at 9 months of the control group | Data of the control group at baseline and 9 months are collected and analyzed.
  Within the control group, prealbumin at 9 months is compared to baseline. In other words, change from baseline prealbumin at 9 months is compared to 0.
Change from Baseline Hemoglobin at 3 months of the treatment group | Data of the treatment group at baseline and 3 months are collected and analyzed.
  Within the treatment group, hemoglobin at 3 months is compared to baseline. In other words, change from baseline hemoglobin at 3 months is compared to 0.
Change from Baseline Hemoglobin at 3 months of the control group | Data of the control group at baseline and 3 months are collected and analyzed.
  Within the control group, hemoglobin at 3 months is compared to baseline. In other words, change from baseline hemoglobin at 3 months compared to 0.
Change from Baseline Hemoglobin at 6 months of the treatment group | Data of the treatment group at baseline and 6 months are collected and analyzed.
  Within the treatment group, hemoglobin at 6 months is compared to baseline. In other words, change from baseline hemoglobin at 6 months is compared to 0.
Change from Baseline Hemoglobin at 6 months of the control group | Data of the control group at baseline and 6 months are collected and analyzed.
  Within the control group, hemoglobin at 6 months is compared to baseline. In other words, change from baseline hemoglobin at 6 months is compared to 0.
Change from Baseline Hemoglobin at 9 months of the treatment group | Data of the treatment group at baseline and 9 months are collected and analyzed.
  Within the treatment group, hemoglobin at 9 months is compared to baseline. In other words, change from baseline hemoglobin at 9 months is compared to 0.
Change from Baseline Hemoglobin at 9 months of the control group | Data of the control group at baseline and 9 months are collected and analyzed.
  Within the control group, hemoglobin at 9 months is compared to baseline. In other words, change from baseline hemoglobin at 9 months is compared to 0.
Change from Baseline Ferritin at 3 months of the treatment group | Data of the treatment group at baseline and 3 months are collected and analyzed.
  Within the treatment group, ferritin at 3 months is compared to baseline. In other words, change from baseline ferritin at 3 months is compared to 0.
Change from Baseline Ferritin at 3 months of the control group | Data of the control group at baseline and 3 months are collected and analyzed.
  Within the control group, ferritin at 3 months is compared to baseline. In other words, change from baseline ferritin at 3 months is compared to 0.
Change from Baseline Ferritin at 6 months of the treatment group | Data of the treatment group at baseline and 6 months are collected and analyzed.
  Within the treatment group, ferritin at 6 months is compared to baseline. In other words, change from baseline ferritin at 6 months is compared to 0.
Change from Baseline Ferritin at 6 months of the control group | Data of the control group at baseline and 6 months are collected and analyzed.
  Within the control group, ferritin at 6 months is compared to baseline. In other words, change from baseline ferritin at 6 months is compared to 0.
Change from Baseline Ferritin at 9 months of the treatment group | Data of the treatment group at baseline and 9 months are collected and analyzed.
  Within the treatment group, ferritin at 9 months is compared to baseline. In other words, change from baseline ferritin at 9 months is compared to 0.
Change from Baseline Ferritin at 9 months of the control group | Data of the control group at baseline and 9 months are collected and analyzed.
  Within the control group, ferritin at 9 months is compared to baseline. In other words, change from baseline ferritin at 9 months is compared to 0.
Change from Baseline Calcium at 3 months of the treatment group | Data of the treatment group at baseline and 3 months are collected and analyzed.
  Within the treatment group, calcium at 3 months is compared to baseline. In other words, change from baseline calcium at 3 months is compared to 0.
Change from Baseline Calcium at 3 months of the control group | Data of the control group at baseline and 3 months are collected and analyzed.
  Within the control group, calcium at 3 months is compared to baseline. In other words, change from baseline calcium at 3 months is compared to 0.
Change from Baseline Calcium at 6 months of the treatment group | Data of the treatment group at baseline and 6 months are collected and analyzed.
  Within the treatment group, calcium at 6 months is compared to baseline. In other words, change from baseline calcium at 6 months is compared to 0.
Change from Baseline Calcium at 6 months of the control group | Data of the control group at baseline and 6 months are collected and analyzed.
  Within the control group, calcium at 6 months is compared to baseline. In other words, change from baseline calcium at 6 months is compared to 0.
Change from Baseline Calcium at 9 months of the treatment group | Data of the treatment group at baseline and 9 months are collected and analyzed.
  Within the treatment group, calcium at 9 months is compared to baseline. In other words, change from baseline calcium at 9 months is compared to 0.
Change from Baseline Calcium at 9 months of the control group | Data of the control group at baseline and 9 months are collected and analyzed.
  Within the control group, calcium at 9 months is compared to baseline. In other words, change from baseline calcium at 9 months is compared to 0.
Change from Baseline Phosphorus at 3 months of the treatment group | Data of the treatment group at baseline and 3 months are collected and analyzed.
  Within the treatment group, phosphorus at 3 months is compared to baseline. In other words, change from baseline phosphorus at 3 months is compared to 0.
Change from Baseline Phosphorus at 3 months of the control group | Data of the control group at baseline and 3 months are collected and analyzed.
  Within the control group, phosphorus at 3 months is compared to baseline. In other words, change from baseline phosphorus at 3 months is compared to 0.
Change from Baseline Phosphorus at 6 months of the treatment group | Data of the treatment group at baseline and 6 months are collected and analyzed.
  Within the treatment group, phosphorus at 6 months is compared to baseline. In other words, change from baseline phosphorus at 6 months is compared to 0.
Change from Baseline Phosphorus at 6 months of the control group | Data of the control group at baseline and 6 months are collected and analyzed.
  Within the control group, phosphorus at 6 months is compared to baseline. In other words, change from baseline phosphorus at 6 months is compared to 0.
Change from Baseline Phosphorus at 9 months of the treatment group | Data of the treatment group at baseline and 9 months are collected and analyzed.
  Within the treatment group, phosphorus at 9 months is compared to baseline. In other words, change from baseline phosphorus at 9 months is compared to 0.
Change from Baseline Phosphorus at 9 months of the control group | Data of the control group at baseline and 9 months are collected and analyzed.
  Within the control group, phosphorus at 9 months is compared to baseline. In other words, change from baseline phosphorus at 9th month is compared to 0.
Change from Baseline 1,25-(OH) 2-D3 at 3 months of the treatment group | Data of the treatment group at baseline and 3 months are collected and analyzed.
  Within the treatment group, 1,25-(OH) 2-D3 at 3 months is compared to baseline. In other words, change from baseline 1,25-(OH) 2-D3 at 3 months is compared to 0.
Change from Baseline 1,25-(OH) 2-D3 at 3 months of the control group | Data of the control group at baseline and 3 months are collected and analyzed.
  Within the control group, 1,25-(OH) 2-D3 at 3 months is compared to baseline. In other words, change from baseline 1,25-(OH) 2-D3 at 3 months is compared to 0.
Change from Baseline 1,25-(OH) 2-D3 at 6 months of the treatment group | Data of the treatment group at baseline and 6 months are collected and analyzed.
  Within the treatment group, 1,25-(OH) 2-D3 at 6 months is compared to baseline. In other words, change from baseline 1,25-(OH) 2-D3 at 6 months is compared to 0.
Change from Baseline 1,25-(OH) 2-D3 at 6 months of the control group | Data of the control group at baseline and 6 months are collected and analyzed.
  Within the control group, 1,25-(OH) 2-D3 at 6 months is compared to baseline. In other words, change from baseline 1,25-(OH) 2-D3 at 6 months is compared to 0.
Change from Baseline 1,25-(OH) 2-D3 at 9 months of the treatment group | Data of the treatment group at baseline and 9 months are collected and analyzed.
  Within the treatment group, 1,25-(OH) 2-D3 at 9 months is compared to baseline. In other words, change from baseline 1,25-(OH) 2-D3 at 9 months is compared to 0.
Change from Baseline 1,25-(OH) 2-D3 at 9 months of the control group | Data of the control group at baseline and 9 months are collected and analyzed.
  Within the control group, 1,25-(OH) 2-D3 at 9 months is compared to baseline. In other words, change from baseline 1,25-(OH) 2-D3 at 9 months is compared to 0.
Change from Baseline Intact Parathyroid Hormone (iPTH) at 3 months of the treatment group | Data of the treatment group at baseline and 3 months are collected and analyzed.
  Within the treatment group, iPTH at 3 months is compared to baseline. In other words, change from baseline iPTH at 3 months is compared to 0.
Change from Baseline iPTH at 3 months of the control group | Data of the control group at baseline and 3 months are collected and analyzed.
  Within the control group, iPTH at 3 months is compared to baseline. In other words, change from baseline iPTH at 3 months is compared to 0.
Change from Baseline iPTH at 6 months of the treatment group | Data of the treatment group at baseline and 6 months are collected and analyzed.
  Within the treatment group, iPTH at 6 months is compared to baseline. In other words, change from baseline iPTH at 6 months is compared to 0.
Change from Baseline iPTH at 6 months of the control group | Data of the control group at baseline and 6 months are collected and analyzed.
  Within the control group, iPTH at 6 months is compared to baseline. In other words, change from baseline iPTH at 6 months is compared to 0.
Change from Baseline iPTH at 9 months of the treatment group | Data of the treatment group at baseline and 9 months are collected and analyzed.
  Within the treatment group, iPTH at 9 months is compared to baseline. In other words, change from baseline iPTH at 9 months is compared to 0.
Change from Baseline iPTH at 9 months of the control group | Data of the control group at baseline and 9 months are collected and analyzed.
  Within the control group, iPTH at 9 months is compared to baseline. In other words, change from baseline iPTH at 9 months is compared to 0.

OTHER OUTCOMES:
Adverse events (death in 9 months) | The mortality of both groups in the 9 observational months are collected.
  The mortality is compared between the treatment group and the control group within 9 months.
Adverse events (cardio-cerebrovascular accidents in 9 months) | The incidence of cardio-cerebrovascular accidents of both groups in the 9 observational months are collected.
  The incidence of cardio-cerebrovascular accidents is compared between the treatment group and the control group within 9 months.
Adverse events (vascular access failure in 9 months） | The incidence of vascular access failure of both groups in the 9 observational months are collected.
  The incidence of vascular access failure is compared between the treatment group and the control group within 9 months.
Drug Safety (liver function-ALT at 9 months) | Data of the both groups at 9 months are collected and analyzed.
  The alanine transaminase(ALT) level at 9 months is compared between the treatment group and the control group.
Drug Safety (liver function-AST at 9 months) | Data of the both groups at 9 months are collected and analyzed.
  The aspartate transaminase(AST) level at 9 months is compared between the treatment group and the control group.
Drug Safety (blood lipid-TG at 9 months) | Data of the both groups at 9 months are collected and analyzed.
  The triglyceride (TG) level at 9 months is compared between the treatment group and the control group.
Drug Safety (blood lipid-TC at 9 months) | Data of the both groups at 9 months are collected and analyzed.
  The total cholesterol (TC) level at 9 months is compared between the treatment group and the control group.
Drug Safety (blood lipid-LDLC at 9 months) | Data of the both groups at 9 months are collected and analyzed.
  The low density lipoprotein cholesterol (LDLC) level at 9 months is compared between the treatment group and the control group.
Drug Safety (blood glucose at 9 months) | Data of the both groups at 9 months are collected and analyzed.
  The random blood glucose level at 9 months is compared between the treatment group and the control group.